CLINICAL TRIAL: NCT06568822
Title: Examining the Relationship Between Physical Activity, Life Satisfaction, and Medication Adherence Outcomes Among Older Turkish Adults
Brief Title: Physical Activity, Life Satisfaction and Medication Adherence in Older Adults
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Deniz Tuncer, Principal Investigator, Bezmialem Vakif University
Other Study IDs: 10/01/2024-136736
Record Dates: First submitted 2024-08-19; First posted 2024-08-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Physical Activity; Life Satisfaction; Medication Adherence; Older Adults
Keywords: Physical Activity; Life Satisfaction; Medication Adherence; Older Adults
MeSH Terms: conditions — Motor Activity; Personal Satisfaction; Medication Adherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older Adults
  Interventions: Other: Asessment; Other: The Physical Activity Scale for the Elderly (PASE); Other: Turkish Version of the Satisfaction with Life Scale (T-SWLS); Other: Modified Morisky Scale (MMS)

INTERVENTIONS:
Other: Asessment — Data prepared by researchers regarding the general characteristics of older adults will be examined.
  Other Names: Sociodemographic Information Form
Other: The Physical Activity Scale for the Elderly (PASE) — PASE will be used to assess the physical activity levels of older adults.
  Other Names: PASE
Other: Turkish Version of the Satisfaction with Life Scale (T-SWLS) — T-SWLS will be used to assess life satisfaction of older adults.
  Other Names: T-SWLS
Other: Modified Morisky Scale (MMS) — MMS will be used to evaluate medication adherence in older adults.
  Other Names: MMS

SUMMARY:
This study will examine the relationships between physical activity, life satisfaction, and medication adherence in elderly individuals with chronic diseases. The research will involve participants aged 65 and above, using the The Physical Activity Scale for the Elderly scale to assess physical activity, the Turkish version of the Satisfaction with Life Scale for life satisfaction, and the Modified Morisky Scale for medication adherence.

DETAILED DESCRIPTION:
The Physical Activity Scale for the Elderly will be used to assess the physical activity levels of geriatric patients. Life satisfaction will be measured using the Turkish version of the Satisfaction with Life Scale, and medication adherence will be evaluated with the Modified Morisky Scale. The data collection will involve forms, including a Sociodemographic Information Form, the Physical Activity Scale for the Elderly, Turkish version of the Satisfaction with Life Scale, and the Modified Morisky Scale, all of which will be digitized using Google Forms. The Google Forms link will then be shared via email by the researchers with individuals who have elderly family members. Before starting to complete the scales with older patients who meet the inclusion and exclusion criteria, they will be informed about the study's purpose, the forms involved, and the time required for completion.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* Voluntarily participating
* Having at least one chronic disease such as hypertension, diabetes mellitus, or hyperlipidemia
* With prescribed medication for the medical treatment of their diagnosed chronic disease

Exclusion Criteria:

* Presence of chronic neurological diseases such as Multiple Sclerosis (MS), Parkinson's Disease, or Amyotrophic Lateral Sclerosis (ALS)
* Any oncological disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults who are prescribed medication due to at least one chronic disease such as hypertension, diabetes mellitus, or hyperlipidemia
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Physical Activity | One Month
  The Physical Activity Scale for Elderly (PASE) will be used to assess the physical activity of elderly individuals. The overall PASE score ranges from 0 to 400 or more, with higher scores indicating better physical activity levels.
Life Satisfaction | One Month
  Turkish version of the Satisfaction with Life Scale (T-SWLS) is a one-dimensional Likert-type scale consisting of 5 questions. The total score of the scale is calculated by adding the scores given to the statements in the scale. The total Turkish version of the SWLS score varies between 5 and 25, and higher scores indicate a better level of life satisfaction.
Medication Adherence | One Month
  The Modified Morisky Scale (MMS) will be used to examine the patient's compliance with treatment by evaluating the motivation and knowledge levels of individuals with chronic diseases regarding pharmacological treatment during long-term treatment. The total score that can be obtained from the scale varies between 0 and 6.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Estebsari F, Dastoorpoor M, Khalifehkandi ZR, Nouri A, Mostafaei D, Hosseini M, Esmaeili R, Aghababaeian H. The Concept of Successful Aging: A Review Article. Curr Aging Sci. 2020;13(1):4-10. doi: 10.2174/1874609812666191023130117. PMID 31657693
- [Background] Barrio-Cortes J, Castano-Reguillo A, Beca-Martinez MT, Bandeira-de Oliveira M, Lopez-Rodriguez C, Jaime-Siso MA. Chronic diseases in the geriatric population: morbidity and use of primary care services according to risk level. BMC Geriatr. 2021 Apr 26;21(1):278. doi: 10.1186/s12877-021-02217-7. PMID 33902470